CLINICAL TRIAL: NCT01845831
Title: Randomized Controlled Trial on the Safety and Efficacy of Sitagliptin Therapy for the Inpatient Management of General Medicine and Surgery Patients With Type 2 Diabetes
Brief Title: Sitagliptin Therapy in Hospitalized Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Temple University (Other); University of Michigan (Other); Ohio University (Other)
Responsible Party: Principal Investigator, Guillermo Umpierrez, Professor of Medicine, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00063642
Record Dates: First submitted 2013-04-30; First posted 2013-05-03 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; DPP4 inhibitors; Sitagliptin; Glargine; RCT; basal insulin; hospital hyperglycemia; inpatient diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Sitagliptin Phosphate; Insulin Glargine; Insulin Aspart; Insulin Lispro; Sitagliptin Phosphate, Metformin Hydrochloride Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Sitagliptin + glargine (Hospital) (Experimental): Sitagliptin and glargine once daily + correction doses of aspart or lispro if needed
  Interventions: Drug: Sitagliptin; Drug: Glargine
- Basal bolus (Hospital) (Active Comparator): Glargine once daily and rapid-acting insulin before meals + correction doses of aspart or lispro if needed
  Interventions: Drug: Basal Bolus
- Metformin and Sitagliptin (Experimental): Patients with HbA1c ≤ 7% will be discharged on the combination of metformin and sitagliptin (Janumet ® 500/50 mg) twice daily for 6 months
  Interventions: Drug: Metformin and Sitagliptin
- Metformin and sitagliptin + glargine 50% (Experimental): Patients with HbA1c between 7% and 9% will be discharged on metformin and sitagliptin (Janumet ® 500/50 mg) twice daily plus glargine insulin (50% of the inpatient glargine dose) for 6 months
  Interventions: Drug: Metformin and Sitagliptin; Drug: Glargine 50%
- Metformin and sitagliptin + glargine 80% (Experimental): Patients with HbA1c > 9% will be discharged on metformin and sitagliptin (Janumet ® 500/50 mg) twice daily plus glargine insulin (80% of the inpatient glargine dose) for 6 months
  Interventions: Drug: Metformin and Sitagliptin; Drug: Glargine 80%

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin will be taken orally at 100 mg or 50 mg once a day per renal function.
  Other Names: Januvia
  Arms: Sitagliptin + glargine (Hospital)
Drug: Basal Bolus — Basal bolus regimen with glargine once daily and rapid-acting insulin (lispro or aspart) before meals + + correction doses of rapid acting insulin if needed
  Other Names: Glargine (Lantus) + aspart (Novolog) or lispro (Humalog)
  Arms: Basal bolus (Hospital)
Drug: Metformin and Sitagliptin — Janumet is a combination of metformin and sitagliptin. Patients with HbA1c ≤ 7% will be discharged on the combination of metformin and sitagliptin (Janumet ® 500/50 mg) twice daily for 6 months.
  Other Names: Janumet
  Arms: Metformin and Sitagliptin; Metformin and sitagliptin + glargine 50%; Metformin and sitagliptin + glargine 80%
Drug: Glargine — Patients with blood glucose between 140-200 mg/dL during hospitalization will receive 0.2 units per kg weight per day.
  Patients with blood glucose between 201-400 mg/dL during hospitalization will receive 0.25 units per kg weight per day.
  Other Names: Lantus
  Arms: Sitagliptin + glargine (Hospital)
Drug: Glargine 50% — Glargine will be prescribed at 50% of daily hospital dose.
  Arms: Metformin and sitagliptin + glargine 50%
Drug: Glargine 80% — Glargine will be prescribed at 80% of daily hospital dose.
  Arms: Metformin and sitagliptin + glargine 80%

SUMMARY:
High blood glucose levels in hospitalized patients with diabetes are associated with increased risk of medical complications and death. Improved glucose control with insulin injections may improve clinical outcome and prevent some of the hospital complications. Glargine (Lantus®) insulin injection is the most common treatment of diabetes in the hospital. Sitagliptin (Januvia®)is effective in lowering blood glucose. In a recent pilot study aiming to determine differences in glycemic control between treatment with sitagliptin (Januvia®) alone or in combination with basal insulin and basal bolus regimen in general medicine and surgery patients with type 2 diabetes (T2D). The investigators found that treatment with sitagliptin alone or in combination with basal insulin resulted in similar glycemic control compared to basal bolus regimen.

The investigators will conduct a prospective RCT aimed to determine the safety and efficacy of sitagliptin therapy for in-hospital and post-discharge management of general medicine and surgical patients with T2D. A total of 280 patients with known history of diabetes will be randomized to receive sitagliptin plus basal (glargine) insulin once daily (group 1), or basal bolus regimen with glargine once daily and aspart or lispro insulin before meals (group 2). If needed, patients in the treatment groups will receive correction doses of rapid-acting insulin in the presence of hyperglycemia (BG > 140 mg/dl). The overall hypothesis is that treatment with sitagliptin in combination with basal insulin in patients with type 2 diabetes will result in a similar improvement in hospital and post-discharge glycemic control and in a lower frequency of hypoglycemic events than treatment with basal bolus insulin regimen with glargine once daily and lispro insulin before meals.

Patients will be recruited at Grady Memorial Hospital, Emory University Hospital, University of Michigan, Ohio State University and Temple University

DETAILED DESCRIPTION:
Specific Aim 1: To determine whether in-hospital glycemic control, as measured by mean daily blood glucose concentration and frequency of hypoglycemic events, is different between treatment with sitagliptin (Januvia®) in combination with basal insulin (glargine) and basal bolus regimen (glargine and rapid-acting insulin analog) in general medicine and surgery patients with T2D. Patients with T2D treated with diet and/or OAD or with low total daily dose insulin therapy (≤0.6 unit/kg/day) will be randomized to receive sitagliptin plus glargine insulin (group 1) or basal bolus regimen with glargine once daily and rapid-acting insulin (lispro or aspart) before meals (group 2). If needed, patients in the 2 treatment groups will receive supplemental (correction) doses of rapid-acting insulin before meals for BG > 140 mg/dl.

Specific Aim 2: To determine the efficacy and safety of an A1C based discharge algorithm in controlling BG after discharge in patients with T2D. Patients who participate in the in-hospital (Aim 1) arm will be invited to enroll in this open label prospective outpatient study. The total duration of the study is 6 months. Patients with HbA1c ≤ 7% will be discharged on the combination of metformin and sitagliptin (Janumet ®) twice daily. Those with HbA1c between 7% and 9% will be discharged on metformin and sitagliptin (Janumet ®) twice daily plus glargine insulin at 50% of the inpatient glargine dose. Those with HbA1c > 9% will be discharged on metformin and sitagliptin (Janumet ®) twice-daily plus glargine insulin at 80% of the inpatient dose.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between the ages of 18 and 80 years admitted to medicine and surgery services.
2. A known history of Type 2 Diabetes > 1 month, receiving either diet alone, oral antidiabetic agents: sulfonylureas and metformin as monotherapy or in combination therapy (excluding DPP-4 inhibitors) or low-dose (≤ 0.6 units/kg/day) insulin therapy.
3. Subjects with a blood glucose >140 mg and < 400 mg/dL at time of randomization without laboratory evidence of diabetic ketoacidosis (serum bicarbonate < 18 mEq/L or positive serum or urinary ketones).

Exclusion Criteria:

1. Age < 18 or > 80 years.
2. Subjects with increased BG concentration, but without a history of diabetes (stress hyperglycemia).
3. Subjects with a history of type 1 diabetes (suggested by BMI < 25 requiring insulin therapy or with a history of diabetic ketoacidosis and hyperosmolar hyperglycemic state, or ketonuria) [46].
4. Treatment with DPP4 inhibitor or Glucagon like peptide 1 (GLP1) analogs during the past 3 months prior to admission.
5. Acute critical illness or coronary artery bypass graft (CABG) surgery expected to require admission to a critical care unit.
6. Subjects with gastrointestinal obstruction or adynamic ileus or those expected to require gastrointestinal suction.
7. Medical or surgical patients expected to be kept NPO for >24-48 hours after admission or after completion of surgical procedure.
8. Patients with clinically relevant pancreatic or gallbladder disease.
9. Patients with acute myocardial infarction, clinically significant hepatic disease or significantly impaired renal function (GFR < 30 ml/min).
10. Treatment with oral or injectable corticosteroid = or > prednisone 5 mg/per day.
11. Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.
12. Female subjects are pregnant or breast feeding at time of enrollment into the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2013-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Umpierrez, MD, Principal Investigator — Emory University SOM
Locations (5):
- United States (5):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - University of Michigan, Ann Arbor, Michigan
  - Ohio State University, Columbus, Ohio
  - Temple University, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Pasquel FJ, Gianchandani R, Rubin DJ, Dungan KM, Anzola I, Gomez PC, Peng L, Hodish I, Bodnar T, Wesorick D, Balakrishnan V, Osei K, Umpierrez GE. Efficacy of sitagliptin for the hospital management of general medicine and surgery patients with type 2 diabetes (Sita-Hospital): a multicentre, prospective, open-label, non-inferiority randomised trial. Lancet Diabetes Endocrinol. 2017 Feb;5(2):125-133. doi: 10.1016/S2213-8587(16)30402-8. Epub 2016 Dec 8. PMID 27964837

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between August 23, 2013 and July 27, 2015.
Pre-assignment Details: Of the 292 subjects who consented for participation, 279 began the inpatient study phase. Two hundred and fifty-three participants began the outpatient study phase.
Groups:
- Sitagliptin + Glargine (Hospital): Inpatient Phase:
  Sitagliptin and glargine once daily + correction doses of aspart or lispro if needed
  Sitagliptin + glargine: Sitagliptin and Glargine once daily + correction doses of rapid acting insulin if needed
- Basal Bolus (Hospital): Inpatient Phase:
  Glargine once daily and rapid-acting insulin before meals + correction doses of aspart or lispro if needed
  Basal Bolus: Basal bolus regimen with glargine once daily and rapid-acting insulin (lispro or aspart) before meals + correction doses of rapid acting insulin if needed
- Metformin and Sitagliptin: Outpatient Phase:
  Patients with HbA1c ≤ 7% during the inpatient phase were discharged on the combination of metformin and sitagliptin (Janumet ® 500/50 mg) twice daily for 6 months
  Metformin and sitagliptin: Patients with HbA1c ≤ 7% were discharged on the combination of metformin and sitagliptin (Janumet ® 500/50 mg) twice daily for 6 months
- Metformin and Sitagliptin + Glargine 50%: Outpatient Phase:
  Patients with HbA1c between 7% and 9% during the inpatient phase were discharged on metformin and sitagliptin (Janumet ® 500/50 mg) twice daily plus glargine insulin (50% of the inpatient glargine dose) for 6 months
  Metformin and sitagliptin + glargine 50%: Patients with HbA1c between 7% and 9% were discharged on metformin and sitagliptin (Janumet ® 500/50 mg) twice daily plus glargine insulin (50% of the inpatient glargine dose) for 6 months
- Metformin and Sitagliptin + Glargine 80%: Outpatient Phase:
  Patients with HbA1c > 9% during the inpatient phase were discharged on metformin and sitagliptin (Janumet ® 500/50 mg) twice daily plus glargine insulin (80% of the inpatient glargine dose) for 6 months
  Metformin and sitagliptin + glargine 80%: Patients with HbA1c > 9% were discharged on metformin and sitagliptin (Janumet ® 500/50 mg) twice daily plus glargine insulin (80% of the inpatient glargine dose) for 6 months
Period: Inpatient Phase
Arm/Group | Sitagliptin + Glargine (Hospital) | Basal Bolus (Hospital) | Metformin and Sitagliptin | Metformin and Sitagliptin + Glargine 50% | Metformin and Sitagliptin + Glargine 80%
Started | 140 | 139 | 0 | 0 | 0
Completed | 139 | 138 | 0 | 0 | 0
Not Completed | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0
Period: Outpatient Phase
Arm/Group | Sitagliptin + Glargine (Hospital) | Basal Bolus (Hospital) | Metformin and Sitagliptin | Metformin and Sitagliptin + Glargine 50% | Metformin and Sitagliptin + Glargine 80%
Started | 0 | 0 | 68 | 98 | 87
Completed | 0 | 0 | 68 | 98 | 87
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The number of participants who received at least one dose of study drug.
Groups:
- Sitagliptin + Glargine (Hospital): Sitagliptin and glargine once daily + correction doses of aspart or lispro if needed
  Sitagliptin + glargine: Sitagliptin and Glargine once daily + correction doses of rapid acting insulin if needed
- Basal Bolus (Hospital): Glargine once daily and rapid-acting insulin before meals + correction doses of aspart or lispro if needed
  Basal Bolus: Basal bolus regimen with glargine once daily and rapid-acting insulin (lispro or aspart) before meals + correction doses of rapid acting insulin if needed
- Total: Total of all reporting groups
Arm/Group | Sitagliptin + Glargine (Hospital) | Basal Bolus (Hospital) | Total
Number analyzed (Participants) | 138 | 139 | 277
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (11.4) | 57.1 (10.4) | 56.9 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 52 | 111
  Male | 79 | 87 | 166
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Race/Ethnicity data were missing for three participants in the Basal/bolus group.
  Participants
    White: number analyzed (Participants) | 138 | 136 | 274
    White | 45 | 44 | 89
    Black: number analyzed (Participants) | 138 | 136 | 274
    Black | 81 | 78 | 159
    Other: number analyzed (Participants) | 138 | 136 | 274
    Other | 12 | 14 | 26

OUTCOME MEASURES:

1. Primary Outcome: Mean Blood Glucose Concentration After First Day of Treatment
Description: The average blood glucose (BG) concentration after the first day of treatment
Time Frame: Duration of Hospitalization (Up to 10 Days)
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Sitagliptin + Glargine (Hospital) | Basal Bolus (Hospital)
Number analyzed (Participants) | 138 | 139
mmol/L | 9.5 (2.7) | 9.4 (2.7)

2. Primary Outcome: Mean Percentage of Blood Glucose Readings Between 3.9 - 7.8 mmol/L
Description: Differences in glycemic control as measured by mean daily blood glucose (BG) concentration between sitagliptin once daily and basal bolus therapy with glargine once daily plus supplemental lispro insulin in hospitalized patients with T2D.
Time Frame: Duration of Hospitalization (Up to 10 Days)
Measure: Mean (Standard Deviation); unit: percentage of blood glucose readings
Groups:
- Basal Bolus (Hospital): Inpatient Phase:
  Glargine once daily and rapid-acting insulin before meals + correction doses of aspart or lispro if needed
  Basal Bolus: Basal bolus regimen with glargine once daily and rapid-acting insulin (lispro or aspart) before meals + + correction doses of rapid acting insulin if needed
Arm/Group | Sitagliptin + Glargine (Hospital) | Basal Bolus (Hospital)
Number analyzed (Participants) | 138 | 139
percentage of blood glucose readings | 30.7 (28.0) | 29.7 (24.4)

3. Primary Outcome: Mean Percentage of Blood Glucose Readings Between 3.9 - 10.0 mmol/L
Description: as for outcome 2
Time Frame: Duration of Hospitalization (Up to 10 Days)
Measure: Mean (Standard Deviation); unit: percentage of blood glucose readings
Arm/Group | Sitagliptin + Glargine (Hospital) | Basal Bolus (Hospital)
Number analyzed (Participants) | 138 | 139
percentage of blood glucose readings | 57.0 (31.5) | 59.6 (30.1)

4. Primary Outcome: Mean Percentage of Blood Glucose Readings Between 5.6 - 7.8 mmol/L
Description: as for outcome 2
Time Frame: Duration of Hospitalization (Up to 10 Days)
Measure: Mean (Standard Deviation); unit: percentage of blood glucose readings
Arm/Group | Sitagliptin + Glargine (Hospital) | Basal Bolus (Hospital)
Number analyzed (Participants) | 138 | 139
percentage of blood glucose readings | 23.3 (21.8) | 23.5 (19.9)

5. Primary Outcome: Mean Percentage of Blood Glucose Readings Greater Than 13.3 mmol/L
Description: as for outcome 2
Time Frame: Duration of Hospitalization (Up to 10 Days)
Measure: Mean (Standard Deviation); unit: percentage of blood glucose readings
Arm/Group | Sitagliptin + Glargine (Hospital) | Basal Bolus (Hospital)
Number analyzed (Participants) | 138 | 139
percentage of blood glucose readings | 14.8 (22.1) | 16.7 (24.1)

6. Primary Outcome: Change in HbA1C
Description: The mean HbA1C measured at 3 months and 6 months post hospitalization. HbA1C is an indicator of diabetes control; below 6.0% is normal, 6.0% to 6.4% indicates prediabetes, and 6.5% or over indicates diabetes.
Time Frame: Post Hospital Discharge Month 3, Month 6
Population: 253 subjects who participated in the inpatient phase and were invited to complete the outpatient phase.
Measure: Mean (Standard Deviation); unit: percent
Groups:
- Metformin and Sitagliptin: Outpatient Phase:
  Patients with HbA1c < 7% during the inpatient phase were discharged on the combination of metformin and sitagliptin (Janumet ® 500/50 mg) twice daily for 6 months
  Metformin and sitagliptin: Patients with HbA1c ≤ 7% were discharged on the combination of metformin and sitagliptin (Janumet ® 500/50 mg) twice daily for 6 months
Arm/Group | Metformin and Sitagliptin | Metformin and Sitagliptin + Glargine 50% | Metformin and Sitagliptin + Glargine 80%
Number analyzed (Participants) | 68 | 98 | 87
percent
  Baseline | 6.3 (.5) | 8.0 (0.6) | 11.3 (1.7)
  Month 3 | 6.3 (.8) | 7.3 (1.1) | 8.0 (1.8)
  Month 6 | 6.2 (1.0) | 7.3 (1.3) | 8.0 (2.0)

7. Secondary Outcome: Number of Participants With a Hypoglycemic Event
Description: The number of participants who had a hypoglycemic event during hospitalization.
Time Frame: Duration of Hospitalization (Up to 10 Days)
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin + Glargine (Hospital) | Basal Bolus (Hospital)
Number analyzed (Participants) | 138 | 139
Participants
  Blood Glucose <3.9 mmol/L | 13 | 17
  Blood Glucose <2.2 mmol/L | 0 | 0

8. Secondary Outcome: Total Daily Insulin Dose
Description: Daily insulin requirement (units per day).
Time Frame: Duration of Hospitalization (Up to 10 Days)
Measure: Mean (Standard Error); unit: units per day
Arm/Group | Sitagliptin + Glargine (Hospital) | Basal Bolus (Hospital)
Number analyzed (Participants) | 138 | 139
units per day | 24.1 (16.2) | 34.0 (20.1)

9. Secondary Outcome: Length of Hospital Stay
Description: Length of hospital stay in days.
Time Frame: Duration of Hospitalization (Up to 10 Days)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Sitagliptin + Glargine (Hospital) | Basal Bolus (Hospital)
Number analyzed (Participants) | 138 | 139
days | 4.0 [3.0 to 8.0] | 4.0 [3.0 to 8.0]

10. Secondary Outcome: Acute Renal Failure Rate
Description: Acute renal failure is defined as a clinical diagnosis of acute renal failure with documented new-onset abnormal renal function (increment > 0.5 mg/dL from baseline).
Time Frame: Duration of Hospitalization (Up to 10 Days)
Measure: Number; unit: participants
Arm/Group | Sitagliptin + Glargine (Hospital) | Basal Bolus (Hospital)
Number analyzed (Participants) | 138 | 139
participants | 7 | 6

11. Secondary Outcome: Hospital Mortality Rate
Description: Mortality is defined as death occurring during admission.
Time Frame: Duration of Hospitalization (Up to 10 Days)
Measure: Number; unit: participants
Arm/Group | Sitagliptin + Glargine (Hospital) | Basal Bolus (Hospital)
Number analyzed (Participants) | 138 | 139
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the duration of the study (2 years) including the inpatient and outpatient phases.
Arm/Group | Sitagliptin + Glargine (Hospital) | Basal Bolus (Hospital)
All-Cause Mortality (participants affected / at risk) | 0/138 | 0/139
Serious Adverse Events (participants affected / at risk) | 10/138 | 9/139
Other Adverse Events (participants affected / at risk) | 2/138 | 1/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin + Glargine (Hospital) (N=138) | Basal Bolus (Hospital) (N=139)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Acute Kidney Injury (Injury, poisoning and procedural complications) | 7 (7) | 6 (6) — Acute renal failure is defined as a clinical diagnosis of acute renal failure with documented new-onset abnormal renal function (increment > 0.5 mg/dL from baseline).
Reoperation (Surgical and medical procedures) | 1 (1) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin + Glargine (Hospital) (N=138) | Basal Bolus (Hospital) (N=139)
Wound Infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
As a single DPP-4 inhibitor, sitagliptin, was used, results cannot be generalized to other incretin-based drugs. Additionally, the proportion of surgical patients was small, and the results may not be generalized to all surgical patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes